CLINICAL TRIAL: NCT03133806
Title: CLASS Canadian Left Atrial Appendage Closure Study
Brief Title: Canadian Left Atrial Appendage Closure Study
Acronym: CLASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-2026
Record Dates: First submitted 2017-04-17; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Left Atrial Appendage; Non-Valvular Atrial Fibrillation
Keywords: Percutaneous Occlusion

STUDY DESIGN:
Intervention Model Description: The study is a multicenter, prospective, single arm design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasept LAA Closure System (Experimental): Interventional percutaneous transcatheter device.
  Interventions: Device: Ultrasept LAA Closure System

INTERVENTIONS:
Device: Ultrasept LAA Closure System — The Ultrasept Left Atrial Appendage Closure System Device is a percutaneous transcatheter device intended to prevent thrombus embolization from the left atrial appendage (LAA) in patients with non-valvular atrial fibrillation.
  Other Names: Ultrasept, Ultrasept LAA Closure Device

SUMMARY:
The purpose of the study is to demonstrate the safety and the rate of closure of the Ultrasept Left Atrial Appendage (LAA) Closure System for the percutaneous occlusion of the left atrial appendage in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
The CLASS study is a multicenter, prospective, single arm trial designed to demonstrate the feasibility and short term efficacy of the Ultrasept Left Atrial Appendage Closure Device. Patients who present or are referred for participation in the study will be evaluated against the inclusion and exclusion criteria. Those meeting the criteria will be given the opportunity to participate. All patients will have protocol-required evaluations at each scheduled follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a documented history of paroxysmal, persistent or permanent non-valvular atrial fibrillation.
* Subject is able to provide informed consent for the procedure.
* Subject is able to be followed for the duration of the study.
* Patient is able to take aspirin and Clopidogrel. Expected duration of dual antiplatelet therapy of 45 days.
* Patient is not able to tolerate or adhere to the requirements of long term anticoagulation therapy.
* Subject has a CHADS score >/= 1.

Exclusion Criteria:

* The patient is known to have an extensive congenital cardiac anomaly which can only be adequately repaired by way of cardiac surgery.
* The patient's size (i.e., too small for TEE probe, catheter size, etc.) or condition (active infection, etc.) would cause the patient to be a poor candidate for cardiac catheterization.
* LAA anatomical exclusion (depth <16mm and/or diameter <11mm).
* Patients with recent myocardial infarction, unstable angina, or decompensated congestive heart failure. (Recent is defined as within 180 days of implant date).
* Patients with any type of serious infection less than one month prior to procedure.
* Patient has demonstrated intracardiac thrombi on echocardiography (especially left atrial or left atrial appendage thrombi).
* Patient is participating in another investigational drug or device study.
* Subject has an implanted atrial septal defect (ASD) device or patent foramen ovale (PFO) device.
* Subject had surgical ASD or PFO repair.
* Subject has a moderate to severe aortic or mitral valve stenosis or regurgitation as assessed by the investigator.
* Subject has a planned ablation procedure for atrial fibrillation within 60 days after the Ultrasept LAA closure device implant.
* Subject has a New York Heart Association (NYHA) grade 4.
* Patient has a left ventricular ejection fraction of 20% or less.
* Patient has a life expectancy of less than one year.
* Subject has had a recent major cardiac surgical procedure (recent is defined as within 180 days of implant date).
* Subject is pregnant, breastfeeding, or desires to become pregnant during their first 180 days post-implant.
* Subject has a medical disorder that would interfere with completion or evaluation of clinical study results (for e.g. uncontrolled hypertension, uncontrolled diabetes, renal failure, in situ inferior vena cava filter).
* Patient has an allergy to Nickel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
Stroke, pericardial effusion, device embolization and device thrombosis | This endpoint will be evaluated at 45 days post-implant.
  The safety endpoints are serious device or procedure-related Adverse Events (SAE) experienced with the Ultrasept Left Atrial Appendage Closure System such as stroke, pericardial effusion requiring treatment, device embolization and device thrombosis.
Peri-device leak rate | This endpoint will be evaluated at 45 days post-implant.
  The efficacy endpoint is completed LAA closure (residual leak < 3 mm) as demonstrated by transesophageal echocardiogram (TEE).

CONTACTS AND LOCATIONS:
Overall Officials: Reda Ibrahim, MD, Principal Investigator — Montreal Heart Institute; Jean-Bernard Masson, MD FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Josep Rodés-Cabau, MD, Principal Investigator — Quebec Heart & Lung Institute Laval University
Locations (1):
- Quebec Heart & Lung Institute Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No